CLINICAL TRIAL: NCT03836404
Title: Pre-market, Multi-center, National, Open-label, Single-arm Study to Evaluate the Safety and Performance of a Class III Medical Device (GreenBone Implant) for Iliac Crest Reconstruction Following Bone Graft Harvesting for Pelvic Fusion
Brief Title: Pre-market Study to Evaluate Safety and Performance of GreenBone Implant
Acronym: GreenBric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GreenBone Ortho S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GB-01-18; NCT03541343 (obsolete NCT alias)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Bone Substitutes
Keywords: Bone substitute; Bone regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iliac Crest reconstruction surgery (Experimental): The patients in the study group will be surgically treated and the GreenBone bone substitute will be implanted
  Interventions: Device: Iliac crest reconstruction surgery

INTERVENTIONS:
Device: Iliac crest reconstruction surgery — When autologous bone graft is needed for the treatment of non-unions or bone defects, is harvested from the pelvic iliac crest. Harvested tricortical graft blocks are used to facilitate fusion of joints (ie pubis symphysis, sacroiliac joint), to structurally support metaphyseal areas of articular impaction injuries and to fill in metaphyseal bone voids. The GreenBone device, with its inherent physical and biomimic properties, possesses similar structural properties to bone, thus, being the ideal material to be used for the treatment of the bone defect (3- 4cm) induced from the harvested tricortical iliac crest, restoring therefore the pelvic anatomy and minimising the risk of chronic pain, haematoma formation and herniation of the abdominal contents.

SUMMARY:
Multi-center, prospective, open-label, single-arm, first-in-human clinical investigation. The patient enrollment will be as follow: initial 5 patients enrolled at PI site. The other remaining patients will be enrolled in the three sites only after positive evaluation of the 3 months Follow Up (FU) interim report analysis by Data Safety Monitoring Board (DSMB). The Patients enrolled in this clinical investigation will undergo a scheduled surgery aiming to reconstruct iliac crest bone defect using GreenBone Implant. After surgery, the Patients will be monitored at pre-scheduled visits up to 6 months. The FU will be extended at 12 months only in case of no complete healing and/or in case of no resolved SAE at the 6 months FU visit. Adverse events, pain, quality of life and X-ray will be evaluated at scheduled follow-up visits. An independent DSMB will review the safety reports at regular intervals and Serious Adverse Events (SAE) as soon as reported, to protect Patients participating in the study. As specified before, an adaptive interim analysis will be performed when at least 5 Patients will have completed the 3 month follow up visit, (V5). The DSMB will review the results of the interim analysis with respect to the primary endpoint (safety) in order to continue the study up to 15 Patients.

DETAILED DESCRIPTION:
This is a pre-market multi-centre, national, open label, single-arm, study to evaluate the safety and performance of a Class III medical device (GreenBone Implant) for iliac crest reconstruction following bone graft harvesting for pelvic fusion. During pelvic fusion a considerable part of the iliac crest is removed and it is used as autologous bone graft for the fusion of the pubis symphysis. The bone defect that is formed in the iliac crest is usually filled with bone obtained from the cows (bovine xenograft) and or human donors (allograft). This carries the risk of transferring disease from animals and/or humans to the patient; there is also a risk of host local allergic reaction. Bone substitutes are devoid of the above risks and therefore they could be used alternatively to xenografts and allografts.

GreenBone is a ceramic resorbable bone scaffold that has very similar structure to bone. It can be produced in large quantities, shaped easily and sterilised without losing its properties. Consequently, it is an ideal substitute that could be used to fill bone defects. This study will assess the safety of using GreenBone to reconstruct iliac crest defects. Moreover it will assess its capacity of promoting new bone formation. The investigators will recruit 15 patients who will undergo pelvic fusion and instead of bovine xenograft the investigators will use the GreenBone implant for the iliac crest reconstruction.

Patients will be followed up for 6 months in total. Safety will be evaluated by monitoring local and potential systemic reactions; its bone forming capacity will also be assessed by its integration into the iliac crest.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Patients.
2. Patients aged ≥ 18 and ≤ 70 years old.
3. Patients requiring iliac crest reconstruction secondary to pelvic fusion.
4. Patients understanding the nature of the study and providing their informed consent to participation.
5. Patients willing and able to attend the visits and procedures foreseen by study protocol.

Exclusion Criteria:

1. Patients with bone infections at the time of enrolment.
2. Patients with bone malignant tumor(s) at the time of enrolment.
3. Patients who have been treated with chemotherapy or radiotherapy within 12 months before the study enrolment.
4. Patients with concomitant infectious systemic diseases at the time of enrolment.
5. Patients with known inflammatory systemic diseases at the time of enrolment.
6. Patients with concomitant myeloproliferative disorders at the time of enrolment.
7. Patients currently treated with systemic immunosuppressive agents, including steroids.
8. Patients with active autoimmune disease.
9. Patients with coagulopathy or bleeding disorders.
10. Patients who have received a previous treatment of bone substitution in the same anatomical site.
11. Patients with known or suspected allergy or hypersensitivity to the GreenBone Implant components.
12. Patients who are participating or have participated in any other conflicting studies within the 30 days before the study enrolment. (This does not include patients who have taken part in other non-conflicting non-interventional or observational studies.

    These patients may still be eligible).
13. Pregnant women and/or women that intend to be pregnant within 6 or 12 months from surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation assessed by Evaluation of adverse events rate | Overall study period up to 6 months
  Evaluation of adverse events rate during the study period. All adverse occurrences (serious/non-serious or device related/non-device related) will be recorded prospectively, categorized and evaluated for causality using defined criteria.

SECONDARY OUTCOMES:
Device Implant Technical Success | At the end of surgical procedure (visit 2, 1 day)
  Technical Success, defined as successful delivery of the bone substitute in the target defect bone evaluated at V2 (at surgical procedure);
Bone regeneration evaluation | At the end of visits 3, 4, 5, 6, 7 (respectively performed 1, 2, 3, 6, 12 months after the surgery, each visit is 1 day)
  Evaluation of the bone regeneration in the area of intervention, by means of X-ray and/or CT examination by a radiologist, on visit V3, V4, V5, V6, V7; X-ray scoring systems have been implemented according to the criteria proposed by Lane and Sandhu (bone formation, union and remodeling) (Lane 1987)
Quality of Life evaluation | At screening visit (V1) and at the end of visits 3, 4, 5, 6, 7 (respectively performed 1, 2, 3, 6, 12 months after the surgery, each visit is 1 day)
  Evaluation of Quality of Life by means of a validated EuroQol questionnaire administered at every visit from V1 to V6/V7 (excluding visit 2) (Price 1983)
Evaluation of Pain | between 1 and 6 months
  Evaluation of degree of pain perceived by the Patient, by means of a Visual Analogue Score (VAS) that a scale with 10 points, from 0 to 10. 0 indicates "no pain at all" and 10 the "worst pain ever"
Treatment tolerability | At the end of visits 3, 4, 5, 6, 7 (respectively performed 1, 2, 3, 6, 12 months after the surgery, each visit is 1 day)
  Evaluation of global tolerability to treatment of Patient (by the Investigator), through a standardized EuroQol questionnaire, on every visit from V3 to V6/V7
Reinterventions number | between 1 and 6 months
  Evaluation of the number of re-interventions occurring for the Patient throughout the . 6 months observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, MD, Principal Investigator — Leeds Teaching Hospital NHS
Locations (1):
- Department of Trauma and Orthopaedic Surgery, Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided